CLINICAL TRIAL: NCT02291003
Title: Identification of Novel Circadian Biomarkers
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Phyllis Zee, Benjamin and Virginia T. Boshes Professor of Neurology, Northwestern University
Other Study IDs: STU00096215
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Circadian Rhythm Disorders
Keywords: circadian; sleep
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, saliva and skin samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy controls: Healthy controls -observational, no intervention administered.

SUMMARY:
Circadian clocks are not only found in discrete areas of the brain, but are found in virtually every organ in our bodies, including the heart, lungs and immune system. Disruptions in circadian clocks, or chronopathology, may underlie various forms of cardiovascular, pulmonary, and metabolic disorders. Over the past two decades, molecular geneticists have "cracked" the clock to reveal its core biochemical mechanisms evident in organisms from fruit flies to humans. These mechanistic insights have led to the discovery of links between clock function and an ever-expanding array of prevalent diseases, including heart, lung, metabolic and sleep disorders. Yet the prevalence of circadian disruption in these patient populations is unclear because current tests are not easily applied in clinical settings or have yet to be developed. Here the investigators exploit our newfound understanding of clock mechanisms and the development of new genomic technologies to identify novel complements of clock-regulated genes ("signatures") that will reveal the state of the internal biological clock. This approach will allow us to take a genomic snapshot of clock status from a single blood draw, substantially easing the diagnosis of these individuals with evidence of circadian disruption or misalignment, i.e., chronopathology.

DETAILED DESCRIPTION:
Circadian clocks are not only found in discrete areas of the brain, but are found in virtually every organ in our bodies, including the heart, lungs and immune system. Disruptions in circadian clocks, or chronopathology, may underlie various forms of cardiovascular, pulmonary, and metabolic disorders. Over the past two decades, molecular geneticists have "cracked" the clock to reveal its core biochemical mechanisms evident in organisms from fruit flies to humans. These mechanistic insights have led to the discovery of links between clock function and an ever-expanding array of prevalent diseases, including heart, lung, metabolic and sleep disorders. Yet the prevalence of circadian disruption in these patient populations is unclear because current tests are not easily applied in clinical settings or have yet to be developed. Perhaps the major limitation of these techniques is the need for serial sampling over extended periods of at least 24 hours and in some cases longer. The development of an assay from a single blood draw would represent a major step forward, facilitating assessments of circadian disruption in a range of diseases.

An alternative strategy to existing assays is to use genomic microarrays to analyze circadian rhythms. Many studies in a number of organisms as well as multiple organs and tissues have found that substantial fractions of the genome (2-10%) are under robust circadian clock control. Importantly, these hundreds of rhythmic genes exhibit expression peaks at all times throughout the day, presumably reflecting their time-of-day specific functions. Using this as a foundation, Ueda and colleagues proposed an alternative strategy that would allow assessment of circadian time from a single blood draw allowing more routine assessments of circadian clock state. In brief, they identified the complement of rhythmic genes in livers of mice. They then selected a set of approximately 50 genes with unique peak times as "time-indicating genes." They then assessed the transcript levels of these time-indicating genes at a single time of day and found that they could accurately determine the time of day that the liver was taken based on the relative expression levels of the time-indicating genes. These studies provide proof-of-principle for the approach that we propose here. Establishing a molecular assay in humans for circadian rhythms from a single time point will allow us to identify circadian rhythm disorders, and to assess internal biological time to deliver therapies at their most efficacious time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls
* Age 18-60
* Intermediate circadian chronotype as determined by the Horne-Ostberg and Munich questionnaire
* Habitual sleep start times between 9:30pm and 1am
* Habitual sleep duration of 6-9 hours

Exclusion Criteria:

* History or current Diagnostic and Statistical Manual-V major psychiatric disorder
* Use of psychoactive medications
* Beck Depression inventory ≥ 16 indicating possible depression
* A history or current diagnosis of a primary sleep disorder (insomnia, sleep apnea, circadian rhythm sleep disorder, restless legs)
* Shift work or other types of self-imposed irregular sleep/wake cycles
* History of, or concurrent unstable or serious medical illness
* Allergy to heparin
* Blindness or other visual impairment other than glasses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy controls, age 18-60 with habitual sleep
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Circadian gene expression profile | 1 day
  The circadian pattern of gene expression will be determined through collecting saliva and blood at regular intervals over a 24 hour and analyzing with microarrays.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis C Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No